CLINICAL TRIAL: NCT06578208
Title: Comparison of Spinal Manipülasyon by Gender in Patients With Chronic Mechanical Low Back Pain
Brief Title: Comparison of the Effect of Spinal Manipulation by Gender
Acronym: CESMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SEFA HAKTAN HATIK (Other)
Responsible Party: Sponsor-Investigator, SEFA HAKTAN HATIK, Assistant Professor, Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CMT0004
Record Dates: First submitted 2024-08-25; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Mechanical Low Back Pain; Chronic Pain; Gender; Neuromuscular Subluxation of Joint
Keywords: Mechanical low back pain; Spinal manipulation; Gender
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Coitus | interventions — Manipulation, Spinal

STUDY DESIGN:
Intervention Model Description: The study included 62 people diagnosed with mechanical low back pain. These 62 people were divided into two groups as male group (n=31) and female group (n=32). Spinal manipulation was performed in the side lying position twice a week for a total of 4 weeks. The evaluation methods were repeated 3 times: at the beginning, at the end and 1 month after the end of the treatment. The study used various statistical techniques to evaluate data, including Shapiro-Wilks test, Student's t test, Mann Whitney U test, repeated measures analysis of variance, Bonferroni test, Friedman's test, Wilcoxon sign test, Wilcoxon Signed Ranks test, and Chi-square test. These tests were used to compare normally distributed and non-normally distributed parameters, as well as within-group comparisons of parameters, and to determine the period causing the difference. Significance was evaluated at a p<0.05 level.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Male Gruop (Experimental): The patient was placed in the lateral decubitus position by the therapist. The foot was placed on the popliteal fossa of the lower leg while the upper knee was flexed. Once the patient was in this position, the therapist performed high velocity and low amplitude thrusts (HVLA; high velocity - low amplitude) on the vertebra with dysfunction.
  Interventions: Other: Spinal Manipulation
- Female Group (Experimental): The patient was placed in the lateral decubitus position by the therapist. The foot was placed on the popliteal fossa of the lower leg while the upper knee was flexed. Once the patient was in this position, the therapist performed high velocity and low amplitude thrusts (HVLA; high velocity - low amplitude) on the vertebra with dysfunction.
  Interventions: Other: Spinal Manipulation

INTERVENTIONS:
Other: Spinal Manipulation — The patient was placed in the lateral decubitus position by the therapist. The foot was placed on the popliteal fossa of the lower leg while the upper knee was flexed. Once the patient was in this position, the therapist performed high velocity and low amplitude thrusts (HVLA; high velocity - low amplitude) on the vertebra with dysfunction (Fagundes Loss et al., 2020).

SUMMARY:
The purpose of the study was to compare and evaluate the effects of spinal manipulation in patients with chronic mechanical low back pain by gender.

DETAILED DESCRIPTION:
Sixty-two participants with a diagnosis of mechanical low back pain participated in the research. 62 individuals were split into two groups based on gender. These were divided into male (n=31) and female (n=31) groups. For four weeks, spinal manipulation was applied twice a week to both groups. The World Health Organization Quality of Life Assessment Short Form (WHOQOL-Bref) was used to evaluate quality of life; the Pittsburg Sleep Quality Index (PSQI) and McGill Pain Questionnaire were used to evaluate sleep quality; Visual Analog Scale (VAS) was used to evaluate pain; Oswetry Disability Index (ODI) was used to evaluate pain-related disability; and a scale was used to evaluate the treatment quality. Range of motion in the hips and lumbar region was measured with a goniometer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic mechanical low back pain
* Between the ages of 18 and 50
* Read and speak Turkish well enough to give informed consent and follow study instruction
* Being able to come for outpatient manipulation treatment
* Body mass index below 28

Exclusion Criteria:

* Currently involved in a legal proceeding related to back pain for which a workers' compensation claim is pending and have or have applied for permanent disability related to these problems
* Pregnancy
* Having any kind of malignancy
* Having any kind of osteoplastic disorders
* Having osteomyelitis, septic intervertebral discs and TB
* History of a spinal fracture and stenosis
* Inflammatory low back pain
* History of severe osteoporosis
* History of any kind of bleeding disorders
* Taking steroids, anticoagulants, paracetamol, antidepressant drugs or drug-like substances
* Having any orthopedic and/or rheumatologic disease affecting the pelvic region
* Conservative or physical therapy for the lumbar region for the past 6 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients diagnosed with mechanical low back pain were included in the study.
Enrollment: 62 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | This questionnaire was conducted at the beginning of treatment, at the end of treatment (week 8) and 1 month after the end of treatment (week 12).
  The VAS used to assess pain intensity consists of a line 10 centimeters (100 millimeters) long. On the lowest score is the expression "I have no pain", on the highest score is the expression "my pain is the worst it can be" and pain is evaluated according to the score expressed between them. The higher the score, the more severe the pain (Sonmezer et al., 2020).
World Health Organization Quality-of-Life Scale (WHOQOL-BREF) | This questionnaire was conducted at the beginning of treatment, at the end of treatment (week 8) and 1 month after the end of treatment (week 12).
  This questionnaire was used to assess quality of life. It consists of 26 questions and includes the categories of physical, psychological, social relations and environment. The higher the score, the higher the quality of life.
Oswetry Disability Index (ODI) | This questionnaire was conducted at the beginning of treatment, at the end of treatment (week 8) and 1 month after the end of treatment (week 12).
  The ODI is a 10-question questionnaire that assesses the disabling effects of low back pain in people suffering from low back pain. Patients self-administer the questionnaire and it takes 7 to 8 minutes for the examiner to evaluate the results. Each question is scored from 0 to 5 and the total score is expressed as a percentage. The higher the score, the higher the level of disability.
Pittsburgh Sleep Quality Index (PSQI) | This questionnaire was conducted at the beginning of treatment, at the end of treatment (week 8) and 1 month after the end of treatment (week 12).
  The PSQI is an effective questionnaire for assessing sleep quality and patterns in adults. It consists of 7 components and sleep quality is rated as "poor" or "good".
McGill Pain Questionnare (MGPQ) | This questionnaire was conducted at the beginning of treatment, at the end of treatment (week 8) and 1 month after the end of treatment (week 12).
  It is a questionnaire designed to measure the sensory, emotional and other effects of pain along with pain intensity in adults with chronic pain. It consists of 4 sections and includes 78 pain descriptive words. The higher the score, the more intense the pain.
Treatment Satisfaction Score | This questionnaire was conducted at the beginning of treatment, at the end of treatment (week 8) and 1 month after the end of treatment (week 12).
  In order to assess the patients' satisfaction with the treatment, similar to the Visual Analog Scale, the expression "I am not satisfied with this treatment" is written on both ends of a 10 cm line at the point where the zero value is located and the expression "I am very satisfied with this treatment" is written at the point where the ten value is located. The patient is asked to mark his/her opinion about this.
Hip and Lumbal ROM Measurements | This questionnaire was conducted at the beginning of treatment, at the end of treatment (week 8) and 1 month after the end of treatment (week 12).
  Range of motion measurements were performed with a goniometer. For hip flexion, supine position was used; the fixed arm of the goniometer was placed on the horizontal axis of the body and the movable arm was placed on the lateral midline of the thigh and the greater trochanter was used as the pivot point. For hip abduction and adduction in the same position, the anterior superior iliac spine was used as the pivot point and the movable arm was placed on the midline of the femur. For hip rotations, the subject's knee and hip were flexed 90°. The fixed arm was placed above the patella apex and parallel to the anterior superior spine and the measurement was made from there. Lumbar ROM measurement was performed according to the description of Otman and Köse (2013).

CONTACTS AND LOCATIONS:
Overall Officials: SEFA HAKTAN HAKTIK, Study Director — Sinop University
Locations (1):
- Sefa Haktan Hatik, Sinop, Turkey (Türkiye)